CLINICAL TRIAL: NCT04267471
Title: Tai Chi for Patients With Essential Hypertension: Study Protocol of an Open-label Single-center Randomized Controlled Trial
Brief Title: Tai Chi for Patients With Essential Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019KL-001
Record Dates: First submitted 2020-02-09; First posted 2020-02-12 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Hypertension
Keywords: Tai Chi; Hypertension; Randomized Controlled Trial
MeSH Terms: conditions — Hypertension | interventions — Tai Ji; Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tai Chi (Experimental): 3 sessions of Tai Chi per week for 12 weeks
  Interventions: Behavioral: Tai Chi
- Walking (Active Comparator): 3 sessions of walking per week for 12 weeks
  Interventions: Behavioral: Walking
- Waiting-list (No Intervention)

INTERVENTIONS:
Behavioral: Tai Chi — Tai Chi is a traditional Chinese mind-body exercise, which combines deep-breath relaxation and gentle movements in sequence with meditation. Each session of Tai Chi will last 60 minutes, including a 10-minute warm-up, a 40-minute Tai Chi practice and a 10-minute cool-down.
  Other Names: Tai Ji Quan
  Arms: Tai Chi
Behavioral: Walking — Each session of walking will last 60 minutes, including a 10-minute warm-up, a 40-minute walking and a 10-minutes cool-down.
  Arms: Walking

SUMMARY:
Several studies investigating Tai Chi for hypertension have been carried out. However, investigators found the results were in high heterogeneity and poor methodological quality. Thus, investigators intend to provide high quality of the effectiveness and safety of Tai Chi for essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. participants aged between 45 to 80 years;
2. participants diagnosed with mild to moderate hypertension, and meet the diagnostic criteria of mild to moderate hypertension according to 2018 Chinese guidelines for the management of hypertension (140≤SBP≤169 and/or 90≤DBP≤109);
3. participants with or without antihypertensive medication;
4. participants with no regular exercise in the past 3 months;
5. participants willing to comply with the study protocol;
6. participants willing to sign informed consent form.

Exclusion Criteria:

1. participants diagnosed with secondary hypertension or refractory hypertension;
2. participants with severe medical visceral condition and chronic diseases, such as diabetes, epilepsy, severe depression or anxiety, psychosis;
3. participants with severe bone and joint diseases or motor dysfunction limit ability to participant exercise;
4. participants with severe cognitive decline (Mini-Mental State Examination score, ≤ 20)
5. participants with weak muscle, poor balance or limited vision that would impede full participation in the study;
6. patients participate in other clinical trials at the same time.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
average 24-h Systolic Blood Pressure (SBP) | change from baseline to 12 weeks after intervention

SECONDARY OUTCOMES:
average SBP and average Diastolic Blood Pressure (DBP) | baseline, after intervention(12 week), after follow-up(24 week)
  average SBP and average DBP during the daytime and night-time
change of serum concentrations of Nitric Oxide | baseline, after intervention(12 week)
change of serum concentrations of endothelin | baseline, after intervention(12 week)
change of serum concentrations of thromboxane A2 | baseline, after intervention(12 week)
change of serum concentrations of vascular endothelial growth factor | baseline, after intervention(12 week)
blood pressure measured at home with an upper arm electronic sphygmomanometer | baseline, after intervention(12 week), after follow-up(24 week)
Medical Outcomes Study 36-Item Short Form | baseline, after intervention(12 week)
  This scale contains eight dimensions (physical function, role physical, bodily pain, general health, vitality, social function, role emotional, mental health) and two summary components (physical and mental), with score from 0 to 100. High scores indicate a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Youping Liu, PhD, Study Chair — Chengdu University of Traditional Chinese Medicine
Locations (1):
- Affiliated Hospital of Chengdu University of Traditional Chinese Medicine (Sichuan Provincial Hospital of Traditional Chinese Medicine), Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li Y, Zhong D, Dong C, Shi L, Zheng Y, Liu Y, Li Q, Zheng H, Li J, Liu T, Jin R. The effectiveness and safety of Tai Chi for patients with essential hypertension: study protocol for an open-label single-center randomized controlled trial. BMC Complement Med Ther. 2021 Jan 7;21(1):23. doi: 10.1186/s12906-020-03192-z. PMID 33413354